CLINICAL TRIAL: NCT00460330
Title: The Value of Real-Time Polymerase Chain Reaction (RT-PCR) Assay, Galactomannan and β-D-Glucan Detection (GM/G-Test) for Diagnosis of Invasive Fungal Infection (IFI) in Chinese Patients After Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Evaluate Three Methods for Diagnosis of Invasive Fungal Infection in Chinese Patients After HSCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Other Study IDs: HXJ-DFI-001
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2007-04-13 (Estimated); Status verified 2007-04

CONDITIONS: Invasive Fungal Infection; Aspergillosis; Fungemia; Hematopoietic Stem Cell Transplantation
Keywords: diagnosis; galactomannan; glucan; real-time PCR; invasive fungal infection; aspergillosis; Chinese patients
MeSH Terms: conditions — Invasive Fungal Infections; Aspergillosis; Fungemia; Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess the cut-off value of GM/G test in Chinese patients after hematopoietic stem cell transplantation, and evaluate GM/G test and real-time PCR for diagnosis of IFI in Chinese patients.

DETAILED DESCRIPTION:
Invasive fungal infection is one of the major complications of HSCT recipients, and the incidence is increased rapidly in recent years. IFI also commonly occurs in Chinese HSCT recipients, and there is no formal report on the mortality and morbidity of IFI in Chinese patients, so this study could supply these data.

Galactomannan(GM) is a cell wall component of aspergillus only, which is released to the blood stream when the aspergillus grows. While the β-D-glucan(BG) is in the most fungal cell wall, and the high level of BG in body fluid is also an evidence of fungal infection. In this study, the serum level of GM and BG would be detected by the commercial available kit.

We will assess the cut-off value of GM/G test by proven/probable IFI patients and negative controls. Then, we could calculate the sensitivity, specificity, positive and negative predict value of the GM/G test. Meanwhile, we may find out the genus of the fungus by comparison of the two methods. For example, both positive of GM and G-test may suggest that the pathogen is Aspergillus, while the positive G-test and negative GM-test implies the Candida may be the pathogen.

RT-PCR is also a helpful method for the IFI diagnosis, which is more sensitive than GM and G-test and encompassing multiple fungal genera. The small-subunit rRNA gene sequence is relatively conserved among members of fungal kingdom, including the Aspergillus and Candida species, the dimorphic fungi, the agents of zygomycosis, and Pneumocystis. So we will amplify that part of DNA and using gene specific probe to detect whether the sample is positive for fungus or not. Until now, there is no report about real-time PCR assay for diagnosis of IFI in Chinese HSCT recipients, so we want to carry out this study. At the same time, the result of real-time PCR assay could help us to estimate the coincidence of GM and G-test with the IFI patients.

After performing the above three diagnostic test, we could identify the HSCT recipients whether they have the IFI more accurately, so that we could evaluate the antifungal therapy and find out the risk factors for IFI in those patients more accurately.

ELIGIBILITY:
Inclusion Criteria:

* Persistent fever(>38.0℃) after three days broad-spectrum anti-bacteria or virus therapy
* Chinese patients after hematopoietic stem cell transplantation

Exclusion Criteria:

* Severe hemolysis patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2007-04; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Jun Huang, Professor, Principal Investigator — Peking University Institute of hematology
Locations (1):
- Institute of Hematology, the People's Hospital, Peking University, Beijing, China